CLINICAL TRIAL: NCT01912183
Title: Family-centred E-health in Pediatric Weight Management: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Katherine Morrison, Associate Professor, Department of Pediatrics, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEH - 126534
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Pediatric Obesity
Keywords: pediatric obesity; e-learning; personal health record; personal electronic device; pilot
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitoring device in PHR (Active Comparator): Both groups will receive routine clinical care in the pediatric weight management program at McMaster Children's Hospital. Children/youth in both groups will receive a physical activity and sleep monitor and access to their PHR. The Active Comparator group will not receive any feedback or communication outside of clinic visits from the clinical team regarding their goal progress.
  Interventions: Behavioral: Monitoring device in PHR; Device: Physical activity and sleep monitor; Other: PHR
- Communication through PHR outside clinic (Experimental): Both groups will receive routine clinical care in the pediatric weight management program at McMaster Children's Hospital. Children/youth in both groups will receive a physical activity and sleep monitor and access to their PHR. The experimental group will receive regular communication with /access to the clinical team through a secure portal within the PHR(i.e. 2 way communication, weekly feedback to the families on their goal progress).
  Interventions: Behavioral: Communication through PHR outside clinic; Device: Physical activity and sleep monitor; Other: PHR

INTERVENTIONS:
Behavioral: Communication through PHR outside clinic
  Other Names: Communication with clinic staff through PHR
  Arms: Communication through PHR outside clinic
Behavioral: Monitoring device in PHR
  Arms: Monitoring device in PHR
Device: Physical activity and sleep monitor
Other: PHR — Access to their PHR

SUMMARY:
This is a pilot study to examine the feasibility of implementing an objective physical activity and sleep monitoring tool into a pediatric weight management program in conjunction with a personal health record (PHR) for children and their families. This feasibility study is intended to provide proof of concept in the incorporation of monitoring devices within the PHR for pediatric patients and their families. Additionally, the investigators will examine whether the PHR helps to empower pediatric patients, their families and the health care team to more effectively monitor the patient's behavior change. Participants will be randomized to receive, or not receive, augmented communication with the health care team between clinical in person visits.

DETAILED DESCRIPTION:
Lifestyle behaviour changes represent the foundation of pediatric weight management and are usually promoted through individual and/or group-based counseling to encourage the adoption and maintenance of health lifestyle behaviours including nutritional intake, sleep and physical activity. Consensus on the need for comprehensive, behavioural interventions exists, but the nature of these interventions vary considerably. The intensity of the intervention (i.e. number of contact hours) may be a key determinant of efficacy, but little detail on the characteristic of these contact hours for optimal delivery is currently available.

In this proof of concept study, we will evaluate the enhancement of behavioural change strategies utilizing technology that provides direct feedback on behaviour change. These devices will be incorporated into a PHR and supplemented with a related e-learning module.

This study will examine the feasibility and perceived usefulness of incorporation of a personal electronic device to encourage behaviour change in children and youth enrolled in a weight management program. We intend to incorporate this device within an established PHR and supplement with evidence-based e-learning.

This is a prospective, randomized pilot study of children and youth (ages 5-17 years) enrolled in a multidisciplinary pediatric weight management program (at McMaster Children's Hospital) for 4 months. This pilot study will include 10 children/youth and parent dyads from each of 3 age groups: 5-9 years, 10-13 years and 14-17 years. All families will utilize a personal electronic device that they can utilize with the individualized PHR. Participants will be randomized to receive, or not receive, regular communication with and access to the clinical team outside of their routine clinical visits, this will occur through a secure portal in the PHR.

ELIGIBILITY:
Inclusion Criteria:

* children/youth between the ages of 5-17 years
* enrolled in pediatric weight management program at McMaster Children's Hospital
* provide informed written assent (child/youth)
* provision of informed written consent (parent/caregiver)

Exclusion Criteria:

* no access to internet/home computer

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Feasibility | 4 months
  Feasibility of the use of personal electronic devices for monitoring behavioural change in response to goal setting through a PHR will be evaluated and compared between the two groups by comparing: 1) percent of consenting families who successfully access the PHR, and 2) percent of children/youth who upload physical activity and sleep data for at least 4/7 days and 75% of weeks of the study.

SECONDARY OUTCOMES:
Acceptability of the personal electronic device and PHR | 2 and 4 months
  Acceptability of the device to the family unit will be evaluated by collating the: 1) number of days per month the family uploads physical activity or sleep information, 2) number of times the family (in the randomized intervention group)interacts with the clinical team through the PHR and 3) number of times over the 4 month period that the family reviews the e-learning module.
  Acceptability of the device and PHR to the child and parent will be ascertained separately via standardized questionnaire at 2 and 4 months after randomization.
Acceptability of goal monitoring | 4 months
  Acceptability of the method of monitoring goal achievement to the clinic staff will be evaluated by questionnaire at the end of the study.
Feasibility of the utilization of the PHR and personal electronic device | 4 months
  Feasibility of the utilization of the PHR and personal electronic device will be measured by examining the percent of eligible, consecutive clinic patients who agree to take part in the study.
Health education | 4 months
  The Health Education Impact Questionnaire (heIQ) will be administered to evaluate the impact of the health education intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Morrison, MD, FRCPC, Principal Investigator — McMaster University/McMaster Children's Hospital
Locations (1):
- Pediatric Weight Management Clinic - McMaster Children's Hospital, Hamilton, Ontario, Canada